CLINICAL TRIAL: NCT01009203
Title: A Phase II Study of Temsirolimus (Torisel®) and Erlotinib (Tarceva®) in Platinum-Refractory or -Ineligible, Advanced, Squamous Cell Carcinoma of the Head and Neck
Brief Title: Temsirolimus (Torisel®) and Erlotinib (Tarceva®) in Platinum-Refractory/Ineligible, Advanced, Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: High patient withdrawal rate
Sponsor: New Mexico Cancer Research Alliance (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST OSI4641s; OSI4641s (Other: Genentech, Inc); NCI-2011-02948 (Registry Identifier: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-07

CONDITIONS: Squamous Cell Carcinoma
Keywords: squamous cell carcinoma; head; neck; aerodigestive
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Erlotinib Hydrochloride; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temsirolimus and Erlotinib (Experimental): Erlotinib (Tarceva) at 150 mg by mouth daily + Temsirolimus (Torisel) at 15 mg intravenously weekly. Each cycle is comprised of 28 days
  Interventions: Drug: Erlotinib; Drug: Temsirolimus

INTERVENTIONS:
Drug: Erlotinib — Treatment will continue until disease progression, unacceptable toxicity, or withdrawal of informed consent.
  Other Names: Tarceva; OSI-774
Drug: Temsirolimus — In the absence of Grade 3 or higher toxicity, a single, intra-patient dose increase of temsirolims to 20 mg intravenously weekly is permitted after the first 28 day cycle. Treatment will continue until disease progression, unacceptable toxicity, or withdrawal of informed consent.
  Other Names: Torisel; CCI-779

SUMMARY:
The primary hypothesis of this study is that the addition of mammalian target of rapamycin (mTOR) blockade to conventional epidermal growth factor receptor (EGFR) blockade will result in synergistic clinical activity in Squamous Cell Carcinoma of the Head and Neck (SCCHN), consistent with preclinical xenograft data. Patients will be treated with the combination of temsirolimus and erlotinib, at the previously established Maximal Tolerated Dose (MTD). The primary signal of efficacy will be progression free survival (PFS), anticipating that PFS will be prolonged compared to historical PFS in SCCHN patients treated with erlotinib or cetuximab monotherapy.

DETAILED DESCRIPTION:
This is a phase II, multicenter, single arm, open-label study. Thirty-seven patients with advanced, platinum-refractory or platinum-ineligible squamous cell carcinoma of the head and neck will be sequentially enrolled to a single treatment arm. Patients will be treated with continuous, 28-day cycles of 150 mg of erlotinib by mouth daily and 15 mg of temsirolimus intervenously weekly. In the absence of grade 3 or higher toxicity in the first cycle, a single, intra-patient dose increase to 20 mg temsirolimus will be permitted.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed squamous cell carcinoma of the head and neck, from any primary site. Nasopharyngeal carcinoma, World Health Organization (WHO) Grade I, will be included.
2. Advanced disease, fulfilling one of the criteria defined below:

   * Incurable disease as assessed by surgical or radiation oncology
   * Metastatic (M1) disease
   * Persistent or progressive disease following curative-intent radiation, and not a candidate for surgical salvage due to incurability or morbidity
3. Platinum-refractory or platinum-ineligible, fulfilling one of the criteria defined below:

   * disease progression during or after 4-6 cycles of platinum-containing therapy in the advanced setting
   * disease progression within 6 months of curative-intent treatment, which included platinum-based chemotherapy
   * ineligible for platinum-containing therapy, in the opinion of the medical oncologist, due to medical comorbidities or unacceptable risk for toxicity
   * patient refuses platinum-containing therapy
4. Measurable disease based on response evaluation criteria in solid tumors (RECIST)

   - disease in previously irradiated sites is considered measurable if there has been unequivocal progression of the lesion after radiotherapy, or the lesion contains residual carcinoma by biopsy more than 6 weeks after completion of radiotherapy
5. Easter Cooperative Oncology Group (ECOG) performance status 0-2 at time of informed consent
6. Adequate hematologic reserve and organ function

   * Absolute neutrophil count > 1200/µl
   * Platelet count > 100,000/µl
   * Renal function: Serum Creatinine ≤ 1.5x upper limit of normal (ULN)
   * Liver function: Total bilirubin ≤ 1.5x ULN, Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5x ULN
7. Able to provide written, voluntary consent
8. Patients with reproductive potential must use an effective contraceptive method.
9. Male or female, age ≥ 18 years
10. Life expectancy ≥ 12 weeks

Exclusion Criteria:

1. Nasopharyngeal primary site, if WHO grade II or III
2. Prior treatment blocking the epidermal growth factor receptor (EGFR), in the advanced disease setting
3. Prior treatment blocking EGFR in the curative-intent setting, if delivered in the previous 6 months
4. Prior treatment with a drug blocking the mammalian target of rapamycin (mTOR)
5. Sensitivity to temsirolimus or erlotinib
6. Uncontrolled metastatic disease of the central nervous system
7. Radiotherapy within the 2 weeks before Cycle 1' Day 1
8. Surgery within the 2 weeks before Cycle 1' Day 1
9. Pregnant or lactating females
10. Myocardial infarction or ischemia within the 6 months preceding study treatment
11. Any co morbid condition that' in the view of the attending physician' renders the patient at high risk from treatment complications
12. No other concurrent, investigational anti-neoplastic agent will be permitted
13. History of prior malignancy within the prior five years, with the exception of non-melanoma carcinomas of the skin, and carcinoma in situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-12; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Homan Fekrazad, MD, Principal Investigator — University of New Mexico Cancer Center
Locations (2):
- United States (2):
  - University of New Mexico Cancer Center @ Lovelace Medical Center, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico

REFERENCES:
- [Result] Bauman JE, Arias-Pulido H, Lee SJ, Fekrazad MH, Ozawa H, Fertig E, Howard J, Bishop J, Wang H, Olson GT, Spafford MJ, Jones DV, Chung CH. A phase II study of temsirolimus and erlotinib in patients with recurrent and/or metastatic, platinum-refractory head and neck squamous cell carcinoma. Oral Oncol. 2013 May;49(5):461-7. doi: 10.1016/j.oraloncology.2012.12.016. Epub 2013 Feb 4. PMID 23384718

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: December, 2009 - March, 2011
Groups:
- Erlotinib and Temsirolimus: Erlotinib at 150 mg by mouth daily + Temsirolimus at 15 mg intravenously weekly. Each cycle is comprised of 28 days.
Period: Overall Study
Arm/Group | Erlotinib and Temsirolimus
Started | 13
Received Treatment | 12 (One patient withdrew consent before treatment started.)
Completed | 6
Not Completed | 7
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 5
Not completed — Treatment-unrelated death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Erlotinib and Temsirolimus
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 61.5 [45 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: The time from treatment initiation to disease progression or death by any cause. Progression is evaluated according to modified Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.0). Target lesions are assessed by computerized tomography (CT) or magnetic resonance imaging (MRI): Progressive Disease (PD), 20% increase in the sum of the longest diameter of target lesions, or unequivocal progression of existing non-target lesion, the appearance of new lesions, death due to disease without prior objective documentation of progression, or global deterioration in health status attributable to disease requiring a change in therapy without objective evidence of progression.
Time Frame: 3 years
Measure: Median (Full Range); unit: Months
Arm/Group | Erlotinib and Temsirolimus
Number analyzed (Participants) | 12
Months | 1.9 [0.6 to 7.4]

2. Secondary Outcome: Toxicity Profile
Description: Toxicities (i.e. Adverse Events) are evaluated prior to each treatment and during any clinical visit. Toxicity will be evaluated per National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), version 3.0. The number of patients affected by adverse events of grade 3 or higher will be reported.
Time Frame: 3 years
Population: Participants who received t least one dose of on-study treatment
Measure: Number; unit: participants
Arm/Group | Erlotinib and Temsirolimus
Number analyzed (Participants) | 12
participants
  Diarrhea | 2
  Facial/neck edema | 1
  Laryngeal edema | 1
  Asthenia | 5
  Peritonitis / infection | 2
  Anorexia | 1
  Elevated triglycerides | 1
  Aspiration pneumonia | 1
  Dyspnea | 3
  Hypoxia | 1

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Tumor response is evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.0). Target lesions are assessed by computerized tomography (CT) or magnetic resonance imaging (MRI:) Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions. Overall response rate (ORR) is the sum of the percentages of patients achieving complete and partial responses
Time Frame: 3 years
Population: Participants evaluable for response
Measure: Number; unit: percentage of evaluable participants
Arm/Group | Erlotinib and Temsirolimus
Number analyzed (Participants) | 9
percentage of evaluable participants
  Complete response (CR) | 0
  Partial response (PR) | 11.1
  Overall response rate (CR + PR) | 11.1

4. Secondary Outcome: Overall Survival (OS)
Description: The time from treatment initiation to death by any cause
Time Frame: 3 years
Measure: Median (Full Range); unit: months
Arm/Group | Erlotinib and Temsirolimus
Number analyzed (Participants) | 12
months | 4 [0.6 to 20.2]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Erlotinib and Temsirolimus
Serious Adverse Events (participants affected / at risk) | 4/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib and Temsirolimus (N=12)
Device related infection (Infections and infestations) | 1 (1)
Cerebrovascular Ischemia (Nervous system disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib and Temsirolimus (N=12)
Rhinitis (Runny nose) (General disorders) | 1 (2)
Leukocytes decreased (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Decreased lymphocytes) (Blood and lymphatic system disorders) | 1 (1)
Neutrophils decreased (Blood and lymphatic system disorders) | 2 (2)
Platelets decreased (Blood and lymphatic system disorders) | 3 (4)
Hypotension (Low blood pressure) (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 10 (20)
Fever (General disorders) | 2 (3)
Weight loss (General disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1 (1)
Fibrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Induration (Hardening of the skin) (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Itching) (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 7 (16)
Wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 1 (2)
Hypothyroidism (Low thyroid function) (Endocrine disorders) | 1 (1)
Anorexia (Loss of appetite) (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 3 (5)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (10)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Heartburn) (Gastrointestinal disorders) | 1 (1)
Dysphagia (Difficulty swallowing) (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Inflammation of the mouth) (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 5 (8)
Taste alteration (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Gingival infection (Gum infection) (Infections and infestations) | 3 (3)
Edema limbs (General disorders) | 2 (2)
Edema: head and neck (General disorders) | 4 (10)
Alkaline phosphatase increased (Investigations) | 1 (1)
Hemoglobin decreased (Investigations) | 2 (2)
Hypercholesterolemia (High cholesterol levels) (Investigations) | 2 (2)
Hyperglycemia (High blood sugar levels) (Investigations) | 3 (3)
Hypertriglyceridemia (High triglyceride levels) (Investigations) | 2 (2)
Hypoalbuminemia (Low albumin levels) (Investigations) | 2 (2)
Hypocalcemia (Low calcium levels) (Investigations) | 2 (2)
Hypokalemia (Low potassium levels) (Investigations) | 4 (6)
Hypomagnesemia (Low magnesium levels) (Investigations) | 3 (3)
Hyponatremia (Low sodium levels) (Investigations) | 1 (1)
Hypophosphatemia (Low phosphate levels) (Investigations) | 2 (3)
Myalgia (Muscle pain) (Musculoskeletal and connective tissue disorders) | 1 (1)
Pelvic soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Syncope (Sudden loss of consciousness) (Nervous system disorders) | 1 (2)
Ear, nose and throat examination abnormal (General disorders) | 6 (11)
Patient odor (General disorders) | 1 (1)
Joint pain (General disorders) | 1 (1)
Neck pain (General disorders) | 1 (1)
Oral pain (General disorders) | 1 (1)
Pain in extremity (General disorders) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Pleural effusion (Fluid collection in lung lining) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Lung collapse) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vascular access complication (Clotting) (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No